CLINICAL TRIAL: NCT07158346
Title: A Randomized, Open, Single-dose, Crossover-design, Phase I Study to Evaluate the Pharmacokinetics and Safety After Co-administration of L03RD1 and L03RD2 or Administration of CT-L03 in Healthy Volunteers
Brief Title: Phase I Study to Evaluate the Pharmacokinetics and Safety After Co-administration of L03RD1 and L03RD2 or Administration of CT-L03 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CT-L03-101
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (L03RD1/L03RD2 -> CT-L03) (Experimental): Administration of 1 tablet of L03RD1 and 2 tablets of L03RD2, and taking 14-day wash-out period, and then administration of 1 table of CT-L03
  Interventions: Drug: L03RD1; Drug: L03RD2; Drug: CT-L03
- B (CT-L03 -> L03RD1/L03RD2) (Experimental): Administration of 1 table of CT-L03, and taking 14-day wash-out period, and then administration of 1 tablet of L03RD1 and 2 tablets of L03RD2
  Interventions: Drug: L03RD1; Drug: L03RD2; Drug: CT-L03

INTERVENTIONS:
Drug: L03RD1 — 1 tablet of L03RD1
Drug: L03RD2 — 2 tablets of L03RD2
Drug: CT-L03 — 1 tablet of CT-L03

SUMMARY:
This is a randomized, open, single-dose, crossover-design, phase I study to evaluate the pharmacokinetics and safety after co-administration of L03RD1 and L03RD2 or administration of CT-L03 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subject is between 19 and 55 years of age, inclusive, at the time of screening.
* 2) Subject has a BMI between 18.0 kg/m² and 29.9 kg/m², inclusive, at the time of screening (≥50 kg for males, ≥45 kg for females).
* 3) Subject's seated blood pressure at the time of screening is 90-139mmHg (systolic) and 60-89 mmHg (diastolic), inclusive.
* 4) Subject who do not have clinically significant congenital or chronic diseases and have no pathological symptoms or findings as a result of internal medical examination. (if necessary, electroencephalography, electrocardiogram, chest and stomach endoscopy, or gastrointestinal radiography, etc.)
* 5) Subject who the principal investigator(or the delegated investigator) determines that he/she is suitable as a study subject as a result of tests performed during screening, such as diagnostic studies(e.g., hematology test, blood chemistry test, serology test, urinalysis) and electrocardiogram(ECG) set and conducted according to the characteristics of the investigational product.
* 6) Subject or his or her spouse or partner agrees to use a medically recognized method of contraception* (excluding hormonal agents) to rule out the possibility of pregnancy from the date of first administration of the investigational product until 14 days after the last administration of the investigational product. They also agree not to donate sperm or eggs.
* 7) Subject who after receiving sufficient explanation and understanding of the purpose, content, characteristics of the investigational product, and expected adverse events, have voluntarily decided to participate and provided written consent.

Exclusion Criteria:

* 1) Subject who have taken a drug that induces or inhibits drug metabolizing enzymes (e.g. barbiturates) within 1 month before the start of the study(date of first administration), or if taken a drug that may affect this study within 10 days before the start of the study(date of first administration).
* 2) Participated in another clinical trial or bioequivalence study and received an investigational product within 6 months of first dose of investigational product.
* 3) Donated whole blood within 8 weeks, blood components within 2 weeks, or received a transfusion within 4 weeks of first dose of investigational product.
* 4) Subject with a history of gastrointestinal resection that may affect drug absorption (excluding appendectomy and hernia surgery).
* 5) Subjects who meet any of the following criteria within 1 month prior to the first dose

  * a. Excessive alcohol consumption
  * b. Smoking more than 20 cigarettes per day
* 6) Subjects with any of the following medical conditions

  * a. Known hypersensitivity to the active ingredient or any component of the investigational product
  * b. Heart failure or a history of heart failure
  * c. Active bladder cancer or history of bladder cancer
  * d. Hepatic impairment
  * e. Severe renal impairment
  * f. Uninvestigated macroscopic hematuria
  * g. Diabetic ketoacidosis, diabetic coma or pre-coma, Type 1 diabetes, or Type 2 diabetes
  * h. Severe infections, perioperative conditions, or moderate trauma
  * i. Genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* 7) Subject with a history of clinically significant mental illness.
* 8) Subject who is judged by the principal investigator(or the delegated investigator) to be unsuitable for this clinical trial for reasons other than the above inclusion/exclusion criteria.
* 9) For female subjects, those who are suspected of being pregnant or breastfeeding.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
AUCt | Pre-dose, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 48, 72 and 96 hours
Cmax | Pre-dose, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 48, 72 and 96 hours

SECONDARY OUTCOMES:
AUCinf | Pre-dose, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 48, 72 and 96 hours
  Area under the plasma concentration-time curve from time 0 to infinity
AUCt/AUCinf | Pre-dose, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 48, 72 and 96 hours
Tmax | Pre-dose, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 48, 72 and 96 hours
  Time of peak plasma concentration
t1/2 | Pre-dose, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 48, 72 and 96 hours
  Half-life
CL/F | Pre-dose, 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 48, 72 and 96 hours

CONTACTS AND LOCATIONS:
Locations (1):
- H plus Yangji Hostpital, Seoul, South Korea